CLINICAL TRIAL: NCT02408341
Title: Effect of Intravenous Propofol Anesthesia Induction on Cardiac Function
Brief Title: Propofol Induction's Effect on Cardiac Function
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Suk Yang, MD, PhD, Assistant Professor, Cardiovascular Medicine, Konkuk University Medical Center
Other Study IDs: KonkukUMC-2012-01
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: This Study Was Focused to Evaluate Feasibility of Doppler Tissue Monitoring During the Induction Anesthesia,; and Evaluate Routine Propofol Induction's Effect on Myocardial Tissue Motion, Using Non-invasive Doppler Tissue and 2D Speckle Tracking Imaging.; This is the First Study, to Our Knowledge, Which Has Evaluated the Possible Impact of Propofol Induction on LV Function.
Keywords: Propofol, Induction anesthesia, Doppler tissue imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine clinical practice of induction anesthesia: There was no intervention, just monitoring of clinical routine practice using non-invasive Doppler tissue imaging.

SUMMARY:
Background: Propofol effects dose-dependent myocardial depression, but there is little clinical data available regarding the direct impact of propofol induction on myocardial function.

Objectives: The purpose of this study was to examine the impact of propofol-based anesthesia induction on cardiac function in low-risk patients.

DETAILED DESCRIPTION:
Study population After approval by the institutional ethics committee and written informed consent, we prospectively enrolled adult patients who were scheduled for elective non-cardiac surgery. During the preoperative anesthesia visit, we selected patients with low-risk as indicated by the revised cardiac risk index of 0 and normal LV function (ejection fraction ≥ 60% and septal e' ≥ 8 cm/s). We excluded patients with an arrhythmia, poor lateral axis in supine position, regional wall motion abnormality, or other structural heart diseases. Patients with any of the following conditions were also excluded: unfavorable airway or facemask fit, intractable coughing, hiccups, or hypotension (mean BP < 60 mmHg) requiring IV positive inotropes or vasoconstrictors during the study period.

Anesthesia induction Upon each patient's arrival at the holding area, we placed an 18-gauge IV line in the right forearm vein and administered 10 mL/kg/hour of lactated Ringer's solution, 0.2 mg of glycopyrrolate, and 0.03 mg/kg of midazolam, as a premedication. Once in the operation room, we started to monitor electrocardiography, non-invasive BP, HR, pulse oximeter oxygen saturation, and the bispectral index (BIS). Anaesthesia induction was started in the following manner. Patients took a spontaneous respiration with inspired oxygen (8 L/min) through a transparent facemask and a circulation system with a reservoir bag. Bolus propofol (2.0 mg/kg) was administered intravenously for 10 seconds, after which assisted ventilation followed. After 5 minutes, complete induction was confirmed via a lack of train-of-four response and followed by tracheal intubation for maintenance anesthesia.

Intraoperative transthoracic echocardiography: Imaging After positioning the patient supine on the operation table, serial transthoracic echocardiography was performed with a portable GE Vivid Q platform (General Electric, Milwaukee, WI), before (T0) and 1, 3, and 5 minutes after the propofol bolus injection (T1, T2 and T3, respectively) along with hemodynamic recordings at the same time (BP, HR, and BIS). Two-dimensional imaging of parasternal and apical views and pulsed wave (PW) Doppler imaging of mitral inflow & LV outflow were performed. DTI was recorded at both septal and lateral mitral annulus from the apical 4-chamber view to determine longitudinal endocardial velocities with a sweep of 66.7 mm/s. Each set of images required less than 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Non-cardiac surgery (already assigned)
* Low risk patients (RCRI score 0)
* Normal Left ventricular systolic function (ejection fraction >= 60%)
* Normal diastolic function (septal e' >= 8cm/s)

Exclusion Criteria:

* Poor echocardiographic imaging
* Emergency surgery
* Unstable hemodynamics (needs positive inotropics)
* Unfavorable airway or facemask
* Coughing, Hiccups

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population After approval by the institutional ethics committee and written informed consent, we prospectively enrolled adult patients who were scheduled for elective non-cardiac surgery. During the preoperative anesthesia visit, we selected patients with low-risk as indicated by the revised cardiac risk index of 0 and normal LV function (ejection fraction ≥ 60% and septal e' ≥ 8 cm/s. We excluded patients with an arrhythmia, poor lateral axis in supine position, regional wall motion abnormality, or other structural heart diseases. Patients with any of the following conditions were also excluded: unfavorable airway or facemask fit, intractable coughing, hiccups, or hypotension (mean BP < 60 mmHg) requiring IV positive inotropes or vasoconstrictors during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes of more than 20% difference of Doppler myocardial tissue systolic motion after propofol administration | 1minute, 3 minutes, 5 minutes
  Anesthesia was induced by intravenous propofol (2.0 mg/kg). We measured tissue Doppler-derived indexes of systolic myocardial motion (S') before and then 1, 3, and 5 minutes after propofol administration. We compared the serial changes by repeated measures ANOVA with Bonferroni post-hoc analyses. More than 20% reduction considered clinically relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea